CLINICAL TRIAL: NCT01538160
Title: A Single and Low Dose of Recombinant Factor VIIa in Patients With Severe Factor XI Deficiency Undergoing Surgery
Acronym: rFVIIa
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-11-8657-OS-CTIL
Record Dates: First submitted 2012-01-19; First posted 2012-02-23 (Estimated); Last update posted 2012-02-23 (Estimated); Status verified 2012-02

CONDITIONS: Hemophilia C
Keywords: recombinant factor VIIa; factor XI deficiency
MeSH Terms: conditions — Factor XI Deficiency | interventions — recombinant FVIIa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: recombinant factor VIIa — single dose of 20ug/kg of recombinant factor VIIa along with tranexamic acid of 4 gram a day for 7 days following surgery

SUMMARY:
Lately the investigators found that patients with severe factor XI deficiency and inhibitors could undergo major surgery with a single low dose of recombinant factor VIIa and tranexamic agent. These results encourage us to apply this treatment in clinical trial setting to patients with severe factor XI deficiency undergoing surgery instead of blood product.

DETAILED DESCRIPTION:
Eligible patients will be those with severe factor XI deficiency who agree to participate in the study . The treatment does not apply to patients requiring coronary artery bypass or other vascular surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients with severe factor XI deficiency who will give informed consent to participate in the study

Exclusion Criteria:

* patients with atherosclerosis disease i.e. unstable angina pectoris or recent stroke
* Patients who required aorto-coronary bypass or any vascular surgery

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2012-02; Primary Completion 2015-07 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Improvement in prophylactic treatment by using single and low dose recombinant FVIIa in patients with severe FXI deficiency | 1 week
  End point to be assessed the degree of bleeding following major operation under rFVIIa

CONTACTS AND LOCATIONS:
Locations (3):
- Israel (3):
  - Ophira Salomon, Ramat Gan
  - Sheba Medical Center, Ramat Gan
  - Sheba Medical Center, Tel Hashomer, Ramat-Gan

REFERENCES:
- [Background] Salomon et al presented at ASH 2008 entitled